CLINICAL TRIAL: NCT06546332
Title: Effectiveness and Safety of the KeriFuse® Intramedullary Arthrodesis Implant and Associated Instruments in the Treatment of IP or DIP Arthritis: a Post Market Clinical Follow-up.
Brief Title: Post Market Clinical Follow-Up KeriFuse®
Status: Active, not recruiting | Type: Observational
Sponsor: Keri Medical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A03148-33
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: KeriFuse® — The intramedullary arthrodesis Implant (KeriFuse®) is indicated for consolidation or bone fusion (arthrodesis) of degraded or arthritic distal interphalangeal (DIP) of hand digits or interphalangeal (IP) joint of the hand thumb.

SUMMARY:
The general objective of this study is to evaluate the performances and the safety related to the KeriFuse® intramedullary arthrodesis implant and associated instrumentation used in accordance with their approved labelling and instruction for use. Performance and safety of KeriFuse® intramedullary arthrodesis implant will be established on short and middle-terms in regards to the implant life-cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years,
* Patients that will have a surgery using a KeriFuse® implant in accordance with the approved labelling and IFU.

Exclusion Criteria:

* Pregnant or nursing women,
* Patients with intellectual disabilities who cannot follow the instructions of their surgeon,
* Patients with a contraindication to surgery and more specifically to the implantation of KeriFuse®,
* Patients with acute or chronic infections, local or systemic,
* Patients with sensitivities or allergies to the implant components (Nickel, Titanium).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The intended target population for the KeriFuse® and associated instruments is an adult population requiring a surgical treatment claimed by the device and presenting bone quality deemed satisfactory by the surgeon.
Sampling Method: Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain and radiological assessment | 3 months
  At 3 months postoperatively, the proportion of patients with a pain level ≤ 3 on VAS (ranking from 0 to 10 cm) and with a fused DIP or IP joint (radiological assessment)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Centre de la main du Pays d'Aix, Aix-en-Provence
  - Clinique de la Chataigneraie, Beaumont
  - Centre Ostéo Articulaire Fleming, Bourgoin
  - Clinique Saint François, Nice
  - Clinique Mutualiste Catalane, Perpignan
  - Clinique du Parc, Périgueux